CLINICAL TRIAL: NCT02305420
Title: EmbryoGen/ Blastgen for Couples With Implantation Problems or Previous Miscarriage
Acronym: BlastGen
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: FertilitySA (Industry)
Collaborators: University of Adelaide (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 8114
Record Dates: First submitted 2014-11-27; First posted 2014-12-02 (Estimated); Last update posted 2018-02-19 (Actual); Status verified 2018-02

CONDITIONS: Recurrent Miscarriage; Infertility
MeSH Terms: conditions — Abortion, Habitual; Infertility

STUDY DESIGN:
Intervention Model Description: Randomised control trial comparing EmbryoGen/ BlastGen media use with standard media in IVF
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- EmbryoGen/BlastGen (Experimental): EmbryoGen and BlasGen media containing GM-CSF 2ng/ml will be used in the experimental arm
  The intervention is to use EmbryoGen/BlastGen
  Interventions: Device: EmbryoGen/ BlastGen media
- Control (Active Comparator): Standard Cook sequential media
  Interventions: Device: Standard Cook sequential media

INTERVENTIONS:
Device: EmbryoGen/ BlastGen media — Embryos will be cultured in media containing Gm-CSF (EmbryoGen/ BlastGen media)
  Other Names: GM-CSF containing media
  Arms: EmbryoGen/BlastGen
Device: Standard Cook sequential media — Standard Cook IVF media will be used in the control arm
  Arms: Control

SUMMARY:
EmbryoGen and BlastGen contain the cytokine growth factor Granulocyte-Macrophage Colony-Stimulating Factor (GM-CSF), which has been documented to give significant benefit to this difficult group of patients.

Results showed a highly significant effect of 44% relative improvement in ongoing implantation rate (p=0.001) in women who have previously miscarried (Ziebe et al 2013).

We wish to undertake a randomised Controlled trial to determine if EmbryoGen/BlastGen media improves pregnancy outcomes in women with recurrent implantation failure, recurrent miscarriage and poor embryo development when compared to standard media.

DETAILED DESCRIPTION:
A randomised control pilot study will be undertaken for 100 women who have implantation failure (≥ 2 embryo transfers without a pregnancy) or at least 1 previous miscarriage and are having a further IVF cycle.

At oocyte retrieval each couple will be randomised using numbered envelopes containing pre randomised group allocations by a person uninvolved in the trial to:

1. BlastGen Group (n=50): culturing their embryos in ORIGIO standard, sequential culture mediums for 3 days (EmbryoGen included) then BlastGen media (GM-CSF containing media) for remaining 2 days or
2. Standard Media Group (n=50): culturing their embryos in Cook standard sequential medium for 5 days.

The best single embryo will be transferred on day 5.

The clinical staff and participating couple will be blinded as to whether BlastGen or standard media was used in culture to day 5. Fertility SA embryologists will not be blind as to which study group a couple is in and which media is being used. The embryos will be cultured using the usual methods and lab facilities by Fertility SA's current embryology staff members who will not be blind to the media being used.

Records on the outcome of the oocyte fertilisation, blastocyst development, implantation rate and pregnancy rates will be recorded, as is standard practice. Pregnancy scans will be carried out at 7 and 12 weeks. Live birth outcomes and any congenital anomalies will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* women undertaking an IVF or ICSI cycle

  * aged between 25 and 41 years
  * 2 or more embryos transferred without a positive pregnancy outcome OR a history of at least 1 previous pregnancy loss, OR
  * Poor embryo development (<20% of embryo developing on time at Day 3 or no blastocyst above Grade 2 on Day 5)

Exclusion Criteria:

* male partner requiring surgical retrieval of sperm except in cases of previous vasectomy
* the use of another investigational drug within 30 days
* any severe chronic disease that would significantly influence an IVF cycle
* less than 3 follicles>14mm on ultrasound on the day of HCG trigger

Ages: 25 Years to 41 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2014-11 (Actual); Primary Completion 2017-06 (Actual); Study Completion 2017-06-14 (Actual)

PRIMARY OUTCOMES:
Livebirth >20 weeks | 9 months after closure of trial (18 +9 months)
  Any delivery >20 resulting in a livebirth

SECONDARY OUTCOMES:
Congenital Anomaly Rate | 9 months after closure of trial (18 +9 months)
  number of liveborns with a congenital anomaly
Clinical pregnancy rates at 7 and 12 weeks gestation | 18 months
  Fetal Heart Beat seen on Ultrasound scan at 7 and 12 weeks
Number of embryos reaching blastocyst stage | 18 months
  Number of blastocysts per cycle
Day 3 and day 5 embryo scores | 18 months
  grade of day 3 and day 5 embryos
Cryopreservation outcomes | 18 months
  Number of Frozen blastocysts

CONTACTS AND LOCATIONS:
Locations (1):
- FertilitySA, Adelaide, South Australia, Australia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rose RD, Barry MF, Dunstan EV, Yuen SM, Cameron LP, Knight EJ, Norman RJ, Hull ML. The BlastGen study: a randomized controlled trial of blastocyst media supplemented with granulocyte-macrophage colony-stimulating factor. Reprod Biomed Online. 2020 May;40(5):645-652. doi: 10.1016/j.rbmo.2020.01.011. Epub 2020 Jan 23. PMID 32220517